CLINICAL TRIAL: NCT06147986
Title: A Phase IIa, Dose-Escalation Followed by Randomized, Open-Label, Parallel-Group Study to Evaluate the Efficacy and Safety of Allogeneic Umbilical Cord Mesenchymal Stem Cells As an Add-On Treatment for Acute ST-elevation Myocardial Infarction (STEMI) Patients
Brief Title: Evaluate the Efficacy and Safety of Allogeneic Umbilical Cord Mesenchymal Stem Cells As an Add-On Treatment for Acute ST-elevation Myocardial Infarction (STEMI) Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ever Supreme Bio Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-CMSC01-A1201
Record Dates: First submitted 2023-05-08; First posted 2023-11-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- UMSC01 (Experimental): UMSC01 cells mixed with normal saline will be administered to patients after the onset of diagnosis of ST-elevation Myocardial Infarction.
  Interventions: Biological: Allogeneic umbilical cord mesenchymal stem cells
- standard treatment (Other): Standard-of-care for ST-elevation Myocardial Infarction
  Interventions: Other: Control group

INTERVENTIONS:
Biological: Allogeneic umbilical cord mesenchymal stem cells — UMSC01 cells will be IC infusion followed by IV infusion with 24 months of follow up after treatment.
  Arms: UMSC01
Other: Control group — Standard-of-care for STEMI
  Arms: standard treatment

SUMMARY:
This phase IIa study is to identify the efficacy and safety of IC(intracoronary) and IV(Intravenous) administrations of UMSC01 in patients with STEMI . This product is a new cell therapy product for treating AMI and produced by Ever Supreme Bio Technology Co., Ltd in Taiwan. The previous Phase I, open-label, single arm, single center study was conducted to evaluate the safety and to explore the efficacy of UMSC01 in subjects with STEMI via intracoronary administration followed by intravenous infusion. This first-in-human Phase I study of UMSC01 was completed on August 2nd, 2021. Among 8 subjects enrolled, no subjects experienced treatment-related TEAEs.

DETAILED DESCRIPTION:
This is a two-stage Phase IIa, dose escalation followed by randomized, open-label, controlled with standard treatment, parallel-group study to evaluate the efficacy and safety of allogeneic umbilical cord mesenchymal stem cell, UMSC01, as an add-on treatment in subjects with STEMI. Subjects should present typical ischemic chest pain within 12 hours after symptoms onset and are diagnosed acute STEMI. Subjects should have undergone standard-of-care for STEMI, the immediate reperfusion management should include primary percutaneous coronary intervention (PCI), aspiration thrombectomy, and adjunctive antithrombotic therapy within 12 hours after the onset of symptoms. This study aims to treat eligible subjects with UMSC01 as an add-on stem cell therapy along with standard-of-care for STEMI. The investigational product (IP), UMSC01, will be applied to subjects via intracoronary (IC) infusion on the 4th - 5th day after the onset of the heart attack, followed by intravenous (IV) infusion 2 days after the IC infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects are aged ≥ 20, < 76 years old on date of consent
2. Presence of typical ischemic chest pain within 12 hours after symptoms onset and clinical diagnosis of acute STEMI according to the 2013 American College of Cardiology (ACC) Foundation/ American Heart Association (AHA) guideline for the Management of STEMI
3. Has undergone standard-of-care for STEMI; the immediate reperfusion management should include primary percutaneous coronary intervention (PCI), aspiration thrombectomy and adjunctive antithrombotic therapy within 12 hours after the onset of symptoms
4. Received successful acute reperfusion therapy (residual stenosis visually < 50% and thrombolysis in myocardial infarction flow ≥ 2) with placement of an intracoronary stent and having a patent infarct-related artery suitable for cell infusion to the target area of abnormal wall motion following myocardial infarction
5. Evidence of LVEF ≥ 30% and < 50% diagnosed by echocardiogram
6. Evidence of stable vital signs prior to IC infusion of UMSC01 (Day 1), defined as no clinical significance of abnormal respiration, afebrile as judged by the investigator, systolic pressure ≥ 90 mmHg and < 160 mmHg, heart rate > 50/min and < 110/min
7. Adequate pulmonary function test defined as a force expiratory volume 1 second (FEV1) > 50% predicted and peripheral artery oxygen saturation ≥ 95% at room air
8. Adequate hematopoietic function at the screening and before administration of study medication:

   * Platelets ≥ 100,000 counts/μL.
   * Hemoglobin ≥ 8 g/dL.
   * PT, APTT ≤ 1.5X upper limit of normal (ULN).
9. Has signed and dated informed consent
10. All male subjects and female subjects with child-bearing potential (between puberty and 2 years after menopause) should use appropriate contraception method(s) shown below, for at least 1 year after the last UMSC01 treatment a. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception) b. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment c. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject d. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3): d.1 Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception d.2 Placement of an intrauterine device (IUD) or intrauterine system (IUS) d.3 Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

Exclusion Criteria:

1. With cardiogenic shock (defined as systolic blood pressure <80mmHg requiring vasopressors, intra-aortic balloon pump(IABP) or extracorporeal membrane oxygenation (ECMO)
2. Presence of severe aortic stenosis or regurgitation according to the recommendation of the 2020 ACC/AHA guideline for themanagement of patients with valvular heart disease
3. Presence of severe mitral stenosis or regurgitation according to the recommendation of the 2020 ACC/AHA guideline for the management of patients with valvular heart disease
4. With a need to undergo staged coronary intervention therapy or coronary artery bypass grafting (CABG) surgery
5. Under an immuno-compromised condition, with known clinically significantly autoimmune conditions, or receiving immunosuppressive treatments within 12 weeks prior to the study intervention
6. Presence of any active malignancy that required treatment within 2 years prior to Screening Visit
7. With ongoing or within the past 2 years serious medical conditions (e.g., concurrent illness), other clinically significant cardiovascular diseases, psychiatric condition (e.g., alcoholism, drug abuse), medical history, physical findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the subject
8. With inadequate hepatic and renal function after onset of STEMI: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 4 x upper limit of normal (ULN); estimated glomerular filtration rate (eGFR) < 40 mL/min, calculated by Modification of Diet in Renal Disease equation (MDRD) 175 formula
9. With uncontrolled diabetes mellitus (blood glucose level > 200 mg/dL or HbA1c ≥ 8.5%)
10. Participation in a clinical trial of an investigational product within 3 months prior to Screening Visit
11. Known or suspected hypersensitivity or previous adverse reaction to any ingredients of study product
12. Female subject with child-bearing potential (between puberty and 2 years after menopause) who is pregnant, lactating or has positive urine pregnancy test at Screening Visit
13. Subjects not suitable to participate the trial as judged by the Investigator(s)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2027-06-24 (Estimated); Study Completion 2027-06-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event (AE) as presented by MedDRA coding system | from Day 1 to 1-month follow-up period
  AE incidences up to 1-month
Incidence of Serious adverse event (SAE) as presented by MedDRA coding system | from Day 1 to 1-month follow-up period
  SAE incidences up to 1-month
Incidence of Suspected and unexpected serious adverse reaction (SUSAR) as presented by MedDRA coding system | from Day 1 to 1-month follow-up period
  SUSAR incidences up to 1-month
Cardiopulmonary Exercise Testing (CPET) | from Day 6 to 6-month follow-up period
  Change in peak oxygen consumption (VO2) at the end of maximal exercise over the study period

SECONDARY OUTCOMES:
Percentage of subject with cardiovascular hospitalizations or urgent care/ emergency room visits for heart failure/exacerbation of coronary artery disease (CAD) | from Day 3 to 24-month follow-up period
  The percentage of subject with cardiovascular hospitalizations or urgent care/ emergency room visits for heart failure/exacerbation of coronary artery disease (CAD) over the study period
Percentage of subject with major adverse cardiovascular events (MACE) | from Day 6 to 24-month follow-up period
  The percentage of subject with major adverse cardiovascular events (MACE), including death, recurrent acute myocardial infarction (AMI), stroke, and target vessel revascularization over the study period
Percentage of subject with ventricular tachycardia/ventricular fibrillation (VT/VF) | from Day 6 to 24-month follow-up period
  The percentage of subject with ventricular tachycardia/ventricular fibrillation (VT/VF) over the study period
New York Heart Association (NYHA) Classification | from Day 6 to 24-month follow-up period
  Changes in New York Heart Association (NYHA) classification over the study period
Echocardiography | from Day 6 to 24-month follow-up period
  Changes in echocardiography variables regional left ventricular wall-motion score index (RWMSI) in total score over the study period
Echocardiography | from Day 6 to 24-month follow-up period
  Changes in echocardiography variables left ventricular end-systolic volume (LVESV) in mL over the study period
Echocardiography | from Day 6 to 24-month follow-up period
  Changes in echocardiography variables left ventricular end-diastolic volume (LVEDV) in mL over the study period
Echocardiography | from Day 6 to 24-month follow-up period
  Changes in echocardiography variables left ventricular ejection fraction (LVEF) in % over the study period
Echocardiography | from Day 6 to 24-month follow-up period
  Changes in echocardiography variables stroke volume (SV) in mL over the study period
Echocardiography | from Day 6 to 24-month follow-up period
  Changes in echocardiography variables LV fractional shortening in % over the study period
Cardiopulmonary Exercise Testing (CPET) | from Day 6 to 24-month follow-up period
  Changes in peak oxygen consumption (VO2) at the end of maximal exercise over the study period
Cardiopulmonary Exercise Testing (CPET) | from Day 6 to 24-month follow-up period
  Changes in exercise time (min) at the end of maximal exercise over the study period
Cardiopulmonary Exercise Testing (CPET) | from Day 6 to 24-month follow-up period
  Changes in ventilatory efficiency/carbon dioxide production (VE/VCO2) slope at the end of maximal exercise over the study period
Cardiopulmonary Exercise Testing (CPET) | from Day 6 to 24-month follow-up period
  Changes in peak heart rate at the end of maximal exercise over the study period
6-minute walk distance (6MWD) | from Day 6 to 24-month follow-up period
  Changes in 6-minute walk distance (6MWD) over the study period
Serum level of amino-terminal pro-brain natriuretic peptide (NT pro-BNP) | from Day 6 to 24-month follow-up period
  Changes in serum level of amino-terminal pro-brain natriuretic peptide (NT pro-BNP) over the study period
cardiac enzyme levels | from Day 6 to 1-month follow-up period
  Changes in cardiac enzyme levels including creatinine kinase (CK), creatinine kinase-MB (CK-MB), and troponin I over the study period
Pulmonary function test | from Day 6 to 24-month follow-up period
  Changes in forced expiratory volume (FEV1) will be tested by Spirometry over the study period
Incidence of adverse event (AE) as presented by MedDRA coding system | from Day 3 to 24-month follow-up period
  AE incidences over the study period
Incidence of serious adverse event (SAE) as presented by MedDRA coding system | from Day 3 to 24-month follow-up period
  SAE incidences over the study period
Incidence of suspected and unexpected serious adverse reactions (SUSAR) s presented by MedDRA coding system | from Day 3 to 24-month follow-up period
  Suspected and unexpected serious adverse reactions (SUSAR) incidences over the study period
12-lead ECG Test | from Day 1 to 24-month follow-up period
  Changes in 12-lead electrocardiogram (ECG) parameters in PR, QRS, QT, QTc, and RR intervals over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Woei C Shyu, Study Director — Ever Supreme Bio Technology Co., Ltd.
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: First-in-human pilot trial of combined intracoronary and intravenous mesenchymal stem cell therapy in acute myocardial infarction — https://www.frontiersin.org/articles/10.3389/fcvm.2022.961920/full